CLINICAL TRIAL: NCT04023916
Title: Phase II Study of Sintilimab Plus R-CHOP as the First-line Treatment for DLBCL Patients With TP53 Mutation and PD-L1 Positive.
Brief Title: Sintilimab Plus R-CHOP as the First-line Treatment in Patients With Diffuse Large B-Cell Lymphoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, vice president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2066
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Diffuse Large B-Cell Lymphoma; Sintilimab; TP53 Mutation
Keywords: DLBCL; Sintilimab; R-CHOP; TP53; PD-L1
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab-R-CHOP (Experimental): Participants with previously untreated DLBCL will receive rituximab and CHOP during Cycle 1 (21-day cycle) and Sintilimab, rituximab, and CHOP during Cycles 2-6 (21-day cycle) ,Sintilimab and rituximab during Cycles 6-8 (21-day cycle) , followed by Sintilimab from Cycles 9-14 (8-week cycle) during consolidation treatment.
  Interventions: Drug: Sintilimab-R-CHOP

INTERVENTIONS:
Drug: Sintilimab-R-CHOP — Drug:Sintilimab:
  Sintilimab:200 mg IV on Day 1 Cycles 2-8, during induction treatment, followed by 200 mg IV on Day 1 of Cycles 9-14.
  Drug: Rituximab Rituximab:Participants with previously untreated DLBCL will receive rituximab at a dose of 375 mg/m^2 IV on Day 1 of Cycle 1-8, during induction treatment.
  Drug: Cyclophosphamide Cyclophosphamide will be administered at a dose of 750 mg/m^2 IV on Day 2 of Cycle 1-6, during induction treatment.
  Drug: Doxorubicin Hydrochloride Liposome Injection Doxorubicin Hydrochloride Liposome Injection will be administered at a dose of 35 mg/m^2 IV on Day 2-3 of Cycle 1-6, during induction treatment.
  Drug: Vincristine Vincristine will be administered at a dose of 1.4 mg/m^2 (maximum 2 mg) IV on Day 2 of Cycle 1-6, during induction treatment.
  Drug: Prednisone Prednisone will be administered at a dose of 40 mg/m^2 orally on Days 1-5 of Cycle 1-6, during induction treatment. Prednisolone may be given if prednisone is unavailable.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sintilimab and R-CHOP regimen as the first-line treatment for DLBCL patients with TP53 mutation and PD-L1 positive.

DETAILED DESCRIPTION:
This Phase II, open-label, single-center, non-randomized study will evaluate the safety and efficacy of induction treatment consisting of Sintilimab in combination with Rituximab plus chemotherapy (R-CHOP) as the first-line treatment in participants with DLBCL, followed by consolidation treatment with Sintilimab alone in patients who achieve CR at the end of induction.For safety reasons, the initial enrollment of the first 6 patients in the study will be slow and conduct intensive monitoring for safety. If the dose-limited toxicity event was observed in more than 2 of the first 6 patients and was assessed caused by cumulative exposure to the study drug combination therapy, the trial will be stopped.This study also aim to evaluate the correlation of clinical efficacy to the expression of PD-L1,PD-1,CD3,CD4,CD8,CD56,CD58,β2-MG，HLA-DR/DP/DQ and so on by immunohistochemical techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as diffuse large B-cell Lymphoma with positive CD20 results;
2. Age between 18 to 70 years old;
3. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2;
4. No history of malignant tumors, having no tumor other than DLBCL at the time of enrollment;
5. Life expectancy no less than 6 months;
6. The patient or his/her attorney would be able to provide written consent for necessary examinations or procedures;
7. Ann Arbor stage I~ IV
8. previously untreated advanced DLBCL.
9. At least one bi-dimensionally measurable lesion (greater than [>] 1.5 centimeters in its largest dimension by CT scan or magnetic resonance imaging)
10. Availability of a representative tumor specimen and the corresponding pathology report for retrospective central confirmation of the diagnosis of DLBCL.
11. Agree to remain abstinent or use contraceptive measures.

Exclusion Criteria:

1. History of autologous stem cell transplantation,radiotherapy or chemotherapy.
2. History of other malignant tumors, except skin basal cell carcinoma and in situ cervical cancer;
3. With uncontrolled cardiovascular/ cerebrovascular disease, coagulation disorders, connective tissue disease, severe infectious diseases;
4. Lymphoma originated in the central nervous system;
5. Left ventricular ejection fraction ≦50％;
6. Abnormal lab results in enrollment:Neutrophil count: <1.5*10^9/L；Platelet count <75*10^9/L；AST or ALT >2 times the upper limit of normal level，AKP and total bilirubin >1.5 times the upper limit of normal level;serum creatinine >1.5 times the upper limit of normal level;
7. Other uncontrolled medical conditions which the investigators think might influence the results of the trial;
8. Patients with mental illnesses or other diseases that might not comply with the trial plan;
9. Women during pregnancy or lactation;
10. HIV positive patients;
11. HbsAg (+) patients with HBV DNA(+), can be enrolled only when his/her HBV DNA turns negative; patients with HBsAg(-) HBcAb(+) can be enrolled only when his/her HBV DNA turns negative;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | every 3 months until 30 months after the last patient's enrollment.
  complete remission rate after treated by Sintilimab+ R-CHOP regimen.

SECONDARY OUTCOMES:
overall survival | 30 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause
adverse events | from the date of first cycle of treatment to 30 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.For safety reasons, the initial enrollment of the first 6 patients in the study will be slow and conduct intensive monitoring for safety. the monitoring time window for each patient is 21 days after the first treatment. If the dose-limited toxicity event was observed in more than 2 of the first 6 patients and was assessed by the research team as caused by cumulative exposure to the study drug combination therapy, the trial will be stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No